CLINICAL TRIAL: NCT07147192
Title: Feasibility Study of an Accommodating IOL Design
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: ILK345-E001
Record Dates: First submitted 2025-08-27; First posted 2025-08-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Aphakia
Keywords: Cataract
MeSH Terms: conditions — Aphakia; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Contralateral implantation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- AAL-FAIOL (Experimental): The clouded lens will be removed by phacoemulsification, after which the AAL-FAIOL will be implanted in one eye.
  Interventions: Device: AAL-FAIOL; Procedure: Phacoemulsification
- BAL-FAIOL (Experimental): The clouded lens will be removed by phacoemulsification, after which the BAL-FAIOL will be implanted in one eye.
  Interventions: Device: BAL-FAIOL; Procedure: Phacoemulsification

INTERVENTIONS:
Device: AAL-FAIOL — Intraocular lens (IOL) placed into the lens capsule of the eye during cataract surgery. IOLs are implantable medical devices intended for long-term use over the lifetime of the pseudophakic subject. Laser energy to specified locations can be used to allow a change in power for far distances.
  Arms: AAL-FAIOL
Device: BAL-FAIOL — Intraocular lens (IOL) placed into the lens capsule of the eye during cataract surgery. IOLs are implantable medical devices intended for long-term use over the lifetime of the pseudophakic subject.
  Arms: BAL-FAIOL
Procedure: Phacoemulsification — Cataract surgery technique that uses ultrasound to break up and remove the clouded lens, allowing for intraocular lens (IOL) implantation.

SUMMARY:
The purpose of this clinical study is to assess safety and explore usability and effectiveness of the test product, AAL-FAIOL. This study will be conducted in Central America.

DETAILED DESCRIPTION:
This study will enroll adult subjects who require cataract surgery in both eyes. One eye will receive the AAL-FAIOL and the other eye will receive the BAL-FAIOL. The two eye surgeries will be separated by 14-35 days. Subjects will attend follow up visits for approximately 1 year. If needed, the AAL lens may be adjusted after surgery with a laser to help give the participant better vision.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Informed Consent Form.
* Willing and able to attend all scheduled study visits required per protocol.
* Diagnosed with bilateral cataracts requiring removal by phacoemulsification.
* Preoperative corneal astigmatism equal to or less than 1.50 diopter (D) in both eyes.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Women of childbearing potential who are pregnant, intend to become pregnant during the study, or are breastfeeding.
* Taking medications that could increase risk or may affect accommodation.
* Eye conditions as specified in the protocol, including glaucoma or ocular hypertension.
* Medical conditions that could increase operative risk as specified in the protocol.
* Other protocol-defined exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative ocular adverse events (AEs), including Secondary Surgical Interventions (SSIs) | From Day 0 up to Month 12
  The number of adverse events, including SSI's, will be calculated. An SSI is a subsequent operation performed to address issues or complications arising from a previous surgical procedure. AEs will be collected starting at Day 0 after informed consent. SSIs will be collected starting Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (5):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States
- Clinica 20/20, San José, Costa Rica
- Instituto Espaillat Cabral, Santo Domingo, Dominican Republic
- Centro Panamericano de Ojos / Clinica Lopez Beltran, San Salvador, El Salvador
- Panama Eye Center, Panama City, Panama